CLINICAL TRIAL: NCT03387774
Title: A Phase 3, Open Label, Multicenter, Randomized Controlled Clinical Trial to Evaluate the Efficacy of Ulinastatin in the Reduction of Acute Oral Mucositis Caused by Concurrent Chemoradiotherapy(CCRT) for Patients With Localregionally Advanced Nasopharyngeal Carcinoma (NPC).
Brief Title: Efficacy of Ulinastatin for Reducing Radiation-Induced Oral Mucositis in Nasopharyngeal Carcinoma Patients
Acronym: UTI-RTOM-NPC
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Collaborators: Affiliated Cancer Hospital & Institute of Guangzhou Medical University (Other); First People's Hospital of Foshan (Other); Fifth Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Zhao Chong, Clinical Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UTI-RTOM-NPC
Record Dates: First submitted 2017-12-02; First posted 2018-01-02 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Oral Mucositis (Ulcerative) Due to Radiation
Keywords: Ulinastatin; Radiation-induced acute oral mucositis; Localregionally Advanced Nasopharyngeal Carcinoma; Intensity Modulated Radiation Therapy
MeSH Terms: conditions — Stomatitis; Ulcer | interventions — Cisplatin; Radiotherapy, Intensity-Modulated; urinastatin; Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Concurrent chemoradiotherapy and ulinastatin (Experimental): Concurrent chemoradiotherapy (CCRT) and intravenous drip of ulinastatin, the details are as follows:
  1. Intensity modulated radiation therapy combined with concurrent chemotherapy of cisplatin 100mg/m2 on day 1 and day 22 of RT;
  2. Ulinastatin through intravenous drip at a dose of one hundred thousand units added to 100 ml of 0.9% normal saline, 3 times every radiation day, until the end of radiotherapy.
  Interventions: Drug: Cisplatin; Radiation: Intensity Modulated Radiation Therapy; Drug: Ulinastatin
- Concurrent chemoradiotherapy (Active Comparator): Concurrent chemoradiotherapy (CCRT) alone:
  Intensity modulated radiation therapy combined with concurrent chemotherapy of cisplatin 100mg/m2 on day 1 and day 22 of RT.
  Interventions: Drug: Cisplatin; Radiation: Intensity Modulated Radiation Therapy

INTERVENTIONS:
Drug: Cisplatin — Patients in both arms received concurrent cisplatin chemotherapy:
  100 mg/m² cisplatin given intravenously every 3 weeks on days 1, 22 concurrently with radiotherapy.
  Other Names: DDP
Radiation: Intensity Modulated Radiation Therapy — Patients in both arms received Intensity Modulated Radiation Therapy:
  All target volumes were outlined slice by slice on the axial contrast-enhanced CT with MR fusion images in the treatment planning system. The target volumes were defined in accordance with the International Commission on Radiation Units and Measurements Reports 50 and 62. The prescribed dose was 68-72 Gy to PTVnx (Planning target volume of the primary tumor), 64-68 Gy to GTVnd (Gross tumor volume of the cervical lymph node), 60- 64Gy to PTVnd and PTV1 (Planning target volume 1), and 54-58 Gy to PTV2 (Planning target volume 2) in 30-32 fractions. The details of dose limits for organs at risk were based on the study 0225 from The Radiation Therapy Oncology Group (RTOG 0225).
  Other Names: IMRT
Drug: Ulinastatin — Patients in the experimental group were received ulinastatin:
  Ulinastatin (UTI): ulinastatin was intravenous drip at a dose of one hundred thousand units added to 100 ml of 0.9% normal saline every time, 3 times every radiation day, and until the end of radiotherapy.
  Other Names: UTI for injection
  Arms: Concurrent chemoradiotherapy and ulinastatin

SUMMARY:
This is a phase 3, open-label, multicenter, randomized controlled phase III clinical trial. The purpose of this study is to evaluate the efficacy of ulinastatin, a kind of protease inhibitor, in the treatment of radiation-induced acute oral mucositis in localregionally advanced nasopharyngeal carcinoma(NPC) patients treated with concurrent chemoradiotherapy(CCRT). To Explore a new and efficient way to reduce the incidence and severity of radiation-induced acute oral mucositis.

DETAILED DESCRIPTION:
Radiation-induced acute oral mucositis (RTOM) in Nasopharyngeal Carcinoma (NPC) patients treat with concurrent chemoradiotherapy (CCRT) is common. Currently, there is no effective treatment for RTOM. Ulinastatin, is a kind of natural anti-inflammatory substance. And this substance is insufficient when the body's inflammatory response is strongly. There are a series of studies have confirmed the efficacy and safety of ulinastatin in the treatment of body's inflammatory response. From the observation of our previous clinical practice, we found that ulinastatin can relieve the severity of RTOM. The present study is undertaken to evaluate the efficacy of ulinastatin in the treatment of RTOM in localregionally advanced NPC patients treated with CCRT.

ELIGIBILITY:
Inclusion Criteria:

* Newly histologic diagnosis of nasopharyngeal carcinoma without distant metastasis
* Clinical stage III~IVa( UICC (Union International Against Cancer) /AJCC (American Joint Committee on Cancer) TNM staging system 8th edition)
* Karnofsky Performance Status Scale between 80-100
* WBC count ≥ 4×109/L，neutrophil differential count≥ 1.5×109/L,Hemoglobin ≥ 90g/L， platelet count ≥ 100×109/L
* ALT or AST ≤2.5×ULN,bilirubin ≤2.5×ULN,Serum creatinine ≤1.5×ULN or Serum creatinine clearance≥60ml/min
* Sign the informed consent.

Exclusion Criteria:

* Angle of sexual squamous cell carcinomas and basal cell layout, squamous cell carcinomas
* Younger than 18 years old or older than 70 years old
* Pregnancy or lactation
* Severe cerebrovascular disease/canker/psychosis/uncontrolled diabetes
* Have suffered from other tumor or now suffering from other tumor
* Have suffered from oral diseases or salivary gland diseases or mow suffering from oral diseases or salivary gland diseases
* Refuse to give up smoking/drinking/betel chewing
* suffering from other active infection diseases and in need of treatment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 179 (Actual)
Dates: Start 2018-01-30 (Actual); Primary Completion 2021-12-28 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
Incidence of Severe Acute Oral Mucositis (Grade of CTC-AE ≥ 3) | Up to 19 weeks
  The primary outcome measures planned in the protocol were the incidence of actue oral mucositis grade greater than or equal to 3 using the Common Terminology Criteria for Adverse Events of Version 4.03 (CTCAE 4.03) in the experimental group and control group. CTCAE 4.03 grade 3 = severe pain; interfering with oral; CTCAE 4.03 grade 4 = Life-threatening consequences; urgent intervention indicated; CTCAE 4.03 grade 5 = death. Mucositis will be assessed weely during concurrent chemoradiotherapy (CCRT) for 7 weeks, and assessed once at 1 month after CCRT and 3 months after CCRT, respectively. The whole observation time may up to 19 weeks.

SECONDARY OUTCOMES:
Weeks to Onset of Severe Radiation-Induced Acute Oral Mucositis (Grade of CTCAE ≥ 3) | Up to Week 19
  Weeks to onset is the duration from the start of radiotherapy to the week of first severe oral mucositis occurred. Severe oral mucositis was defined as a Grade 3 or above of Common Terminology Criteria For Adverse Events of Version 4.03 (CTCAE 4.03). CTCAE 4.03 grade 3 = severe pain; interfering with oral; CTCAE 4.03 grade 4 = Life-threatening consequences; urgent intervention indicated; CTCAE 4.03 grade 5 = death. Mucositis will be assessed weekly during concurrent chemoradiotherapy (CCRT) for 7 weeks, and assessed once at 1 month after CCRT and 3 months after CCRT, respectively. Time to onset of severe mucositis will be recorded. The whole observation time may up to 19 weeks.
Oral Assessment Guide (OAG) Score | Up to 19 weeks
  The Oral Assessment Guide (OAG) score is calculated based on the following categories: ability of swallow; the appearance of lips; the appearance of tongue; the appearance of oral mucous membranes; the appearance of gingivae; the appearance of teeth; and the change of voice. There are three grades in every category. The details about Oral Assessment Guide is available in: http://www.rch.org.au/rchcpg/hospital_clinical_guideline_index/Mouth_Care_of_the_paediatric_oncology_patient/. The OAG score will be assessed weekly during concurrent chemoradiotherapy (CCRT) for 7 weeks, and assessed once at 1 month after CCRT and 3 months after CCRT, respectively. The whole observation time may up to 19 weeks.
Oral Mucositis Scores by World Health Organization (WHO) | Up to 19 weeks
  The Oral Mucositis Score of World Health Organization (WHO) was classified based on the changes of patients' oral mucosa and ability to eat, and are classified to 4 grades. WHO scale for oral mucositis (available in: Peterson DE, Boersdoets CB, Bensadoun RJ, et al. Management of oral and gastrointestinal mucosal injury: ESMO Clinical Practice Guidelines for diagnosis, treatment, and follow-up. Annals of Oncology 2015; 26(supply5). https://doi.org/10.1093/annonc/mdv202): Grade 0 = no oral mucositis; Grade 1 = erythema and soreness; Grade 2 = ulcers, able to eat solids; Grade 3 = ulcers, requires liquid diet (due to mucositis); Grade 4 = ulcers, alimentation not possible (due to mucositis). The WHO score will be assessed weekly during concurrent chemoradiotherapy (CCRT) for 7 weeks, and assessed once at 1 month after CCRT and 3 months after CCRT, respectively. The whole observation time may up to 19 weeks.
Rate of Participants With Unplanned Breaks in Radiotherapy | During the 7 weeks for concurrent chemoradiotherapy
  Participants with a duration of 5 days or more without an administration of radiotherapy or who discontinue radiotherapy prior to completion of planned radiotherapy were considered to have an unplanned break in radiotherapy. The rate of unplanned break was calculated for both arms.
Quality of Life with EORTC QLQ-C30 | Up to 19 weeks
  The quality of life for all participants was evaluated according to The European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30) (available in: Grønvold M. EORTC QLQ-C30 Scoring Manual 2014.). The EORTC QLQ-C30 shoule be completed weekly during concurrent chemoradiotherapy (CCRT) for 7 weeks, and assessed once at 1 month after CCRT and 3 months after CCRT, respectively. The whole observation time may up to 19 weeks.
Karnofsky Performance Status Scale | Up to 19 weeks
  The functional status for all participants was assessed according to Karnofsky Performance Status Scale (KPS Scale) (available in: Friendlander AH, Ettinger RL. Karnofsky performance status scale[J]. Special Care in Dentistry, 2009, 29(4):147.). The KPS Scale was range from 0 to 100, and were averagely divided into eleven grades begin with 0. The KPS Scale will be recoreded weekly during concurrent chemoradiotherapy (CCRT) for 7 weeks, and assessed once at 1 month after CCRT and 3 months after CCRT, respectively. The whole observation time may up to 19 weeks.
Numeric Rating Scale for Pain(NRS scale) | Up to 19 weeks
  The pain caused by oral mucositis for all participants was assessed according to Numeric Rating Scale (NRS scale), by which a respondent selects a whole number (0-10 integers) that best reflects the intensity of their pain. And an 11-point scale where 0 indicates no pain and 10 indicates the worst imaginable pain. The scale for each patient was recorded. The NRS scale will be assessed weekly during concurrent chemoradiotherapy (CCRT) for 7 weeks, and assessed once at 1 month after CCRT and 3 months after CCRT, respectively. The whole observation time may up to 19 weeks.
3 Months Overall Response Rate | Assessed at 3 months after concurrent chemoradiotherapy
  Efficacy was estimated according to Response Evaluation Criteria in Solid Tumor version 1.1 (RECIST 1.1) (available in: Watanabe H, Okada M, Kaji Y, et al. New response evaluation criteria in solid tumours-revised RECIST guideline (version 1.1. European Journal of Cancer, 2009, 45(2):228-247.). The efficacy was divided into complete response (CR), partial response (PR), stable disease (SD), and progressive disease (PD). And CR was defined as disappearance of all target lesions, PR was defined as at least a 30% reduction in the sum of the longest diameter of target lesions. Overall response rate (ORR) is the sum rate of patients with CR and PR for the total number of evaluable patients.
The Adverse events Related to Ulinastatin | Up to 19 weeks
  The adverse events related to ulinastatin based on medicine specification of ulinastatin was observed and recorded down according to Common toxicity criteria, version 2.0. (available in: Version CTC, Version CTC, Date P, et al. Common toxicity criteria (ctc) 1999.).

CONTACTS AND LOCATIONS:
Overall Officials: zhao chong, Principal Investigator — Sun Yat-sen University
Locations (1):
- Cancer Center, Sun Yat-sen University, Guangzhou, Guangdong, China

REFERENCES:
- See also: Home Page of Cancer Center, Sun Yat-sen University — http://www.sysucc.org.cn